CLINICAL TRIAL: NCT02055326
Title: Complementary Treatments for Smoking Cessation
Brief Title: Yoga for Men Attempting Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AT003669-02S1
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-01

CONDITIONS: Smoking Cessation
Keywords: Smoking; yoga; men; intervention
MeSH Terms: conditions — Smoking Cessation; Smoking; Multiple Endocrine Neoplasia Type 1 | interventions — Cognitive Behavioral Therapy; Yoga; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental): One-hour sessions of twice weekly yoga for 8 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Smoking Cessation; Behavioral: Yoga
- Health & Wellness (Active Comparator): 8 week program of health & wellness classes, materials and handouts. Topics included healthy eating, cancer prevention and cardiovascular disease prevention.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Smoking Cessation; Behavioral: Health & Wellness

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Smoking Cessation — one hour weekly for 8 weeks. Cognitive behavioral therapy for smoking cessation
Behavioral: Yoga — One hour, twice weekly for 8 weeks of vinyasa yoga
  Arms: Yoga
Behavioral: Health & Wellness — Lectures, handouts and printed materials on general health and wellness topics including healthy eating, cancer prevention and cardiovascular disease prevention.
  Arms: Health & Wellness

SUMMARY:
The purpose of this pilot study is to examine the feasibility and preliminary efficacy of a quit-smoking program that combines behavioral therapy with either yoga, or a health & wellness program that serves as a contact control.

DETAILED DESCRIPTION:
Men enrolled in this pilot will be provided with 8 weeks of cognitive-behavioral therapy for smoking cessation and either 1) a twice-weekly program of yoga, or 2) a health & wellness program that serves as a control for number of contacts and subject burden between study conditions. Qualitative data from open ended surveys and interviews is used to supplement survey data to enhance the investigators understanding of study outcomes. Participant accrual and retention rates, acceptance of randomization, and compliance with study protocols will be examined along with perceptions and beliefs about yoga and its relationship to quitting smoking specifically, and health in general.

ELIGIBILITY:
Inclusion Criteria:

* male
* age 18 -65
* daily smoker, 5 or more cigarettes/day
* generally healthy
* able to exercise safely

Exclusion Criteria:

* female
* hypertension
* current or recent history of medication use for major depression
* participation in yoga classes within the past year
* current or >1 year prior experience with mind/body therapies
* currently participating in regular exercise classes
* currently enrolled in quit smoking program
* currently using quit smoking medications

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-09; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence | 7 days
  7-day point prevalence abstinence was measured at 8 weeks, 3 and 6 months follow up

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700